CLINICAL TRIAL: NCT02628522
Title: A Novel Method for Chronic Anal Fissure Treatment: Adipose Derived Regenerative Cells - A Pilot Study
Brief Title: A Novel Method for Chronic Anal Fissure Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Katarina Andjelkov, Clinical professor, principal investigator, Clinical Centre of Serbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCS-1
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Anal Fissure
Keywords: ADRC; Celution
MeSH Terms: conditions — Fissure in Ano | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRCs therapy (Experimental): Infiltration with 20mL Lidocaine 2% and Epinephrine 1:100 000. Liposuction will be done from the abdomen using Tulip cannulas. Fat will be processed with Celution system.
  Isolated ADRCs will be administered in chronic anal fissures.
  Interventions: Other: ADRCs therapy; Device: Celution; Device: Tulip cannulas; Other: 20mL Lidocaine 2% and Epinephrine 1:100 000

INTERVENTIONS:
Other: ADRCs therapy — Patients with chronic anal fissures will receive one treatment of local injections of fat enriched with adipose derived regenerative cells starting from December 2014.
Device: Celution — Adipose derived regenerative cell isolation
Device: Tulip cannulas — Lipoaspiration
Other: 20mL Lidocaine 2% and Epinephrine 1:100 000 — Infiltration prior to liposuction
  Other Names: Xylocaine 2% and adrenaline 1:100 000

SUMMARY:
Investigators performed a prospective pilot study to test the feasibility and safety of autologous adipose derived regenerative cell (ADRC) transplantation in treatment of anal fissures. The study included 6 patients with chronic anal fissures with symptoms that had an average duration of 24 months. All patients were candidates for surgical treatment as all previous conservative treatments were unsuccessful. The pain level was measured using the VAS scale and was recorded before the treatment and on every consultation following the treatment.

The initial hypothesis is that application of ADRCs may be an alternative to lateral sphincterotomy and a reliable procedure to avoid fecal incontinence.

DETAILED DESCRIPTION:
This prospective pilot study includes 6 patients suffering from chronic anal fissure. All patients were previously treated with different local applications of glyceryl trinitrate or topical Xylocaine gel. Some patients took oral analgesics as a concomitant therapy for additional pain control. None of the patient received neither topical calcium channel blockers nor Botulinum toxin injection due to the unavailability.

The primary outcome measured is "time to complete cessation of anal pain". The secondary outcome includes the healing of chronic anal fissure defined as "time to complete epithelization".

The study was approved by the Ethics Committee of the First Surgical Clinic, Faculty of Medicine, and University of Belgrade. The study was performed in accordance with the Declaration of Helsinki and current Good Clinical Practices. All patients gave the written informed consent prior to the participation.

Physical examination and the detail medical history has been taken by an experienced colorectal surgeon. Pain assessment is quantified using the visual analog scale (VAS) before the treatment and during each postoperative outpatient visit. Bowel continence has been also assessed using Wexner fecal incontinence score prior to the treatment and during each postoperative outpatient visit. The liposuction procedure has been performed performed under the combination of local anesthesia and moderate sedation/general anesthesia. The mixture of 180 mL saline solution, 1mL Epinephrine (1:10,000) and 20 mL of 2% lidocaine is injected in the subcutaneous layer of the abdominal wall to allow the tumescence and to decrease the blood loss. The manual liposuction procedure has been carried out through two or three small incisions using Sforza harvester (Tulip® medical products, San Diego, USA). Approximately 150-200 mL of raw lipoaspirate is obtained from each patient. The harvest site is then covered with a pressure dressing for 10 days to reduce swelling and hematoma. The closed system PureGraft® 250mL (PureGraft®, Solana Beach, California, USA) has been used used to collect the specimen. The specimen is transferred within 15 min to the BelPrime Clinic laboratory where the Celution® 800/CRS system (Cytori Therapeutics, Inc. San Diego, California, USA) is applied to process the lipoaspirate in order to obtain ADRCs. The Celution® 800/CRS system is a closed automated medical device that helps to separate blood and fat. The system will then digests fat using the proprietary enzyme reagent Celase 835/CRS (Cytori Therapeutics, Inc. San Diego, California, USA) to release the stromal vascular fraction (SVF). SVF is subsequently concentrated by a short centrifugation and then automated wash cycles to obtain the ADRC fraction. This 90 to 120-minute process provides approximately 5mL of pellet. A few drops of the obtained pellet were immediately used for cell counting (ChemoMetec A/S DK-3450, Allerod, Denmark).

The second procedure has been performed in lithotomy position. Intravenous prophylactic antibiotic (1gm Metronidazol) are administered. After the careful and gentle anal examination, anal fissure is first curetted using a small size curette. The pellet is divided into two parts. The first 2mL of the pellet is mixed with 8mL of the lipid part of the lipoaspirate purified by Puregraft® 50 system. This solution (10mL) is injected subcutaneously into the edge of the fissure using the criss-cross lattice technique by Tulip® 1,2 mm injector. The rest of the pellet, (approximately 2-5mL), is infiltrated directly into the fissure base (internal anal sphincter) using a 20G needle. No laxatives or stool softener is prescribed. Patients have been discharged from the hospital a few hours after the procedure.

Patients are followed up weekly by telephone interview during the first 2 months, then monthly up to 12 months after the procedure. The outpatient visits are scheduled monthly until 9 months to ensure the healing of anal fissure. Visual analogue scale (VAS) score and Wexner fecal incontinence score [31] are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were adults (>18 years) with chronic (> 8 weeks of conservative therapy) anal fissures

Exclusion Criteria:

* The exclusion criteria were autoimmune diseases, inflammatory bowel disease, presence of malignant or chronic infectious disease, or immunosuppressive therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Time to complete cessation of anal pain | 33 days

SECONDARY OUTCOMES:
Time to complete epithelization | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Andjelkov, MD, PhD, Principal Investigator — Clinical Centre Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Result] Fox A, Tietze PH, Ramakrishnan K. Anorectal conditions: anal fissure and anorectal fistula. FP Essent. 2014 Apr;419:20-7. PMID 24742084
- [Result] Ommer A, Wenger FA, Rolfs T, Walz MK. Continence disorders after anal surgery--a relevant problem? Int J Colorectal Dis. 2008 Nov;23(11):1023-31. doi: 10.1007/s00384-008-0524-y. Epub 2008 Jul 16. PMID 18629515
- [Result] Voswinkel J, Francois S, Simon JM, Benderitter M, Gorin NC, Mohty M, Fouillard L, Chapel A. Use of mesenchymal stem cells (MSC) in chronic inflammatory fistulizing and fibrotic diseases: a comprehensive review. Clin Rev Allergy Immunol. 2013 Oct;45(2):180-92. doi: 10.1007/s12016-012-8347-6. PMID 23296948
- [Result] Borowski DW, Gill TS, Agarwal AK, Bhaskar P. Autologous adipose-tissue derived regenerative cells for the treatment of complex cryptoglandular fistula-in-ano: a report of three cases. BMJ Case Rep. 2012 Nov 9;2012:bcr2012006988. doi: 10.1136/bcr-2012-006988. PMID 23144344
- [Derived] Andjelkov K, Sforza M, Barisic G, Soldatovic I, Hiranyakas A, Krivokapic Z. A novel method for treatment of chronic anal fissure: adipose-derived regenerative cells - a pilot study. Colorectal Dis. 2017 Jun;19(6):570-575. doi: 10.1111/codi.13555. PMID 28574663